CLINICAL TRIAL: NCT06581692
Title: Non-invasive Monitoring of Miscarriage
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2024.354
Record Dates: First submitted 2024-08-23; First posted 2024-09-03 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Miscarriage in First Trimester

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood, Products of conception
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is a routine procedure, no intervention will be provided. — This is a routine procedure, no intervention will be provided.

SUMMARY:
cfDNA is extremely useful to ascertain chromosomal causes of miscarriages at the point of miscarriage diagnosis by a simple blood test. This study aims to determine the level of cell-free DNA (cfDNA) in early pregnancy and compare the results with those of product of conception (POC) testing, in concordance with standard karyotyping.

DETAILED DESCRIPTION:
Pregnancies achieved by assisted reproductive technologies (ART) are closely monitored, therefore miscarriages that occur very early in the pregnancy are frequently meticulously recorded and reported. On the other hand, spontaneous abortion rates among naturally occurring conceptions are notoriously hard to quantify and are often overstated when using criteria from assisted reproductive technologies. Additionally, women who have undergone treatment with ART are a particular population with traits that can make them more vulnerable to spontaneous abortions.

cfDNA would be extremely useful to ascertain chromosomal causes of miscarriages at the point of miscarriage diagnosis by a simple blood test. This study aims to determine the level of cell-free DNA (cfDNA) in early pregnancy and compare the results with those of product of conception (POC) testing, in concordance with standard karyotyping.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years.
2. Women who attend the early pregnancy loss clinic or Patients who receive ART
3. Their partner, the biological father of the pregnancy

Exclusion Criteria:

* History of psychological/ psychiatric problem
* Patient refusal

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Patients will be approached on the day of attending the early pregnancy loss clinic, and given information about the study. Sufficient time will be allowed for consideration before they confirm their decision and sign the consent. For cases with the management of ultrasound-guided manual vacuum aspiration (USG-MVA) or surgical evacuation, their remaining products of gestation will be collected for analysis.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2039-08-31 (Estimated); Study Completion 2039-08-31 (Estimated)

PRIMARY OUTCOMES:
Cell-free DNA (cfDNA) | 15 weeks
  Determine the use of cfDNA to ascertain chromosomal causes of miscarriages

SECONDARY OUTCOMES:
Level of cell-free DNA | 15 weeks
  To determine the level of cell-free DNA (cfDNA) in early pregnancy
Aneuploidy results from product of conception | 15 weeks
  To compare the aneuploidy results from product of conception (POC), in concordance with standard karyotyping.

CONTACTS AND LOCATIONS:
Overall Officials: PUI WAH JACQUELINE CHUNG, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No